CLINICAL TRIAL: NCT01411514
Title: Phase IV Study of Oral Prednisone Taper vs. Placebo Following Intravenous Steroids for the Treatment of Acute Relapses in Multiple Sclerosis Within the Ticino Cohort
Brief Title: Oral Prednisone Taper Versus Placebo for the Treatment of Acute Relapses in Multiple Sclerosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulties to recruit patients
Sponsor: Claudio Gobbi (Other Government)
Collaborators: Ente Ospedaliero Cantonale, Ticino, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Claudio Gobbi, Dr. med., Ospedale Civico, Lugano
Organization: Ospedale Civico, Lugano (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EOC.NC.10.04
Record Dates: First submitted 2011-05-26; First posted 2011-08-08 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing remittent multipse sclerosis; Secondary progressive multiple sclerosis; Clinically isolated syndrome; Primary progressive multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisone (Experimental)
  Interventions: Drug: Prednisone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisone — Tablets, 60 mg od p.o. for 5 days, followed by 40 mg o.d. p.o. for 5 days, 20 mg o.d. p.o. for 5 days, 10 mg o.d. p.o. for 5 days, 5 mg o.d. p.o. for 5 days
  Other Names: Prednison Axapharm
  Arms: Prednisone
Drug: Placebo — Placebo tablets. They will be administered during 25 days
  Other Names: Placebo tablets
  Arms: Placebo

SUMMARY:
The management of MS-patients requires treatment with immune-modifying or immune-suppressive agents to prevent new relapses and progression of disability. Several studies have evaluated the effect of steroid treatment on clinical recovery after an acute relapse. An important unanswered clinical question is, whether or not an oral tapering dose of corticosteroids offers any additional advantage over intravenous methylprednisolone alone in improving neurologic recovery as well as safety and tolerability after a relapse.

This study aims to compare the efficacy, tolerability and safety of tapering doses of oral prednisone and placebo after short-term high-dose i.v. methylprednisolone on the recovery from an acute relapse in patients with clinically isolated syndrome (CIS), relapsing-remitting multiple sclerosis (RR-MS) and primary (PP-MS) or secondary progressive multiple sclerosis (SP-MS) with superimposed relapses.

Patients will be treated during 25 days with de-escaling doses of prednisone or placebo.

The primary analysis will test whether placebo is equivalent to oral prednisone taper on the recovery status as measured by EDSS change from baseline to 3 months after baseline.

DETAILED DESCRIPTION:
The purpose of this double-blind, randomised, placebo-controlled, prospective, parallel group, single centre study is to evaluate the effect of tapering oral doses of prednisone or placebo taken during 25 days following short-term high-dose i.v. methylprednisolone on the outcome of a relapse in patients with CIS; RR-MS, PP-MS or SP-MS with superimposed relapses. The primary objective is to assess and compare the recovery status in both patient groups 3 months after baseline by means of Expanded Disability Status Scale (EDSS). Secondary objectives are the assessments of clinical parameters at the end of oral treatment, 6, 9 months after baseline, of MRI markers, of mental and cognitive status, quality of life and fatigue at the end of oral treatment, 3 and 6 months after baseline in both patient groups.

After standard treatment of an acute clinical relapse with high dose, short term i.v. methyprednisolone patients will be randomised to one of the two treatment arms. Patients allocated to prednisone will be treated with tapering oral doses during 25 days. The initial dose of 60 mg will be reduced twice by 20 mg, than by 10 and 5 mg. Each dose regimen will be taken during 5±2 days. Patients randomised to placebo will receive placebo treatment during 25 days.

ELIGIBILITY:
Inclusion Criteria:

* female or male
* aged between 18 and 80 years;
* with relapsing forms of multiple sclerosis diagnosed according to McDonald's criteria, including RR-MS and relapsing SP-MS, CIS, PP;
* with EDSS score between 0 and 8;
* experiencing an acute relapse with a documented clinical worsening of at least one point of the EDSS scale or a worsening of at least 2 points in one of the EDSS functional systems;
* having agreed to have MRI and having already received at least one enhanced MRI before study procedures without major side effects;
* having agreed to adhere to the study procedures;
* having signed the written informed consent form.

Exclusion Criteria:

* secondary progressive MS without superimposing relapses;
* primary progressive MS without superimposed relapses;
* patients suffering from any clinical condition contraindicated for steroid, in particular

  * Systemic fungal infection
  * Severe osteoporosis
  * Uncontrolled hypertension or congestive heart failure.
  * Existing or previous history of severe affective disorders (especially previous steroid psychosis).
  * Diabetes mellitus
  * History of tuberculosis
  * Glaucoma
  * Previous corticosteroid-induced myopathy
  * Liver failure or cirrhosis
  * Renal insufficiency
  * Active epilepsy
  * Peptic ulceration
  * Fresh intestinal anastomoses
  * Predisposition to thrombophlebitis
  * Abscess or other pyogenic infections
  * Diverticulitis
  * Myasthenia gravis
  * Ocular herpes simplex
  * Hypothyroidism
  * Recent myocardial infarction
  * Kaposi's sarcoma;
* any disease other than multiple sclerosis that would better explain the patient's signs and symptoms;
* women of potential childbearing without active contraceptive methods;
* pregnancy (urine pregnancy test at baseline visit) or breast feeding;
* history of affective disorders;
* history of attempted suicide or current suicidal ideas;
* medical or psychiatric conditions that compromise the ability to give informed consent, to comply with the protocol, or to complete the study;
* inability, in the opinion of the principal investigator or staff, to comply with protocol requirements for the duration of the study;
* known hypersensitivity to prednisone or excipients of the study medications;
* any contraindication for concomitant medications;
* any contraindication for MRI or contrast administration;
* a history of drug abuse in the 6 months prior to screening;
* use of steroids during the previous 30 days (disease-modifying therapies for the treatment of MS are allowed);
* treatment with drugs that might interfere with the evaluation of study drugs during the study protocol (see Section 4.2.2);
* likelihood of requiring treatment during the study period with drugs not permitted by the study protocol;
* participation in an other clinical trial within 30 days prior to entry in this study or current participation in another trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | baseline, 3 months
  The scores of the Expanded Disability Status Scale (EDSS) will be assessed at baseline, defined as start of oral treatment with prednisone or placebo (Day 1), and 3 months after baseline.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | baseline, 25 days (end of treatment)
  the scores of the Expanded Disability Status Scale (EDSS) will be assessed at baseline, at end of treatment, 6, and 9 months after baseline;
Multiple Sclerosis Functional Composite Score (MSFC) | baseline, 25 days (end of treatment)
  the Multiple Sclerosis Functional Composite Score (MSFC) includes the Timed 25 foot-walk-test, the 9 Hole Peg test and Paced Auditorial Addition Test (PASAT)
Gd-enhancing lesions on T1-weighted images | baseline, 25 days (end of treatment)
  the evolution of the number of Gd-enhancing lesions on T1-weighted images will be assessed
number of new T2-hyperintense lesions | baseline, 25 days (end of treatment)
  the evolution of the number of new T2-hyperintense lesions will be assessed
mental status (MUSIC) | baseline, 25 days (end of treatment)
  investigator administered questionnaire
Euroqol-5D (EQ-5D | baseline, 25 days (end of treatment)
  patient reported quality of life
Functional Assessment Multiple Sclerosis (FAMS) | at baseline, 25 days (end of treatment)
  Patient reported outcome
Beck Depression Inventory Second edition (BDI-II) | baseline, 25 days (end of treatment)
  Investigator administered questionnaire
Fatigue Scale for Motor and Cognitive functions (FSMC) | baseline, 25 days (end of treatment)
  Investigator administered questionnaire
Expanded Disability Status Scale (EDSS) | baseline, 6 months
  The scores of the Expanded Disability Status Scale (EDSS) will be assessed at baseline, defined as start of oral treatment with prednisone or placebo (Day 1), and 6 months after baseline.
Expanded Disability Status Scale (EDSS) | baseline, 9 months
  The scores of the Expanded Disability Status Scale (EDSS) will be assessed at baseline, defined as start of oral treatment with prednisone or placebo (Day 1), and 9 months after baseline.
Multiple Sclerosis Functional Composite Score (MSFC) | baseline, 3 months
  the Multiple Sclerosis Functional Composite Score (MSFC) includes the Timed 25 foot-walk-test, the 9 Hole Peg test and Paced Auditorial Addition Test (PASAT)
Multiple Sclerosis Functional Composite Score (MSFC) | baseline, 6 months
  the Multiple Sclerosis Functional Composite Score (MSFC) includes the Timed 25 foot-walk-test, the 9 Hole Peg test and Paced Auditorial Addition Test (PASAT)
Multiple Sclerosis Functional Composite Score (MSFC) | baseline, 9 months
  the Multiple Sclerosis Functional Composite Score (MSFC) includes the Timed 25 foot-walk-test, the 9 Hole Peg test and Paced Auditorial Addition Test (PASAT)
Gd-enhancing lesions on T1-weighted images | baseline, 3 months
  the evolution of the number of Gd-enhancing lesions on T1-weighted images will be assessed
Gd-enhancing lesions on T1-weighted images | baseline, 6 months
  the evolution of the number of Gd-enhancing lesions on T1-weighted images will be assessed
number of new T2-hyperintense lesions | baseline, 3 months
  the evolution of the number of new T2-hyperintense lesions will be assessed
number of new T2-hyperintense lesions | baseline, 6 months
  the evolution of the number of new T2-hyperintense lesions will be assessed
mental status (MUSIC) | baseline, 3 months
  investigator administered questionnaire
mental status (MUSIC) | baseline, 6 months
  investigator administered questionnaire
Euroqol-5D (EQ-5D | baseline, 3 months
  patient reported quality of life
Euroqol-5D (EQ-5D | baseline, 6 months
  patient reported quality of life
Functional Assessment Multiple Sclerosis (FAMS) | at baseline, 3 months
  Patient reported outcome
Functional Assessment Multiple Sclerosis (FAMS) | at baseline, 6 months
  Patient reported outcome
Beck Depression Inventory Second edition (BDI-II) | baseline, 3 months
  Investigator administered questionnaire
Beck Depression Inventory Second edition (BDI-II) | baseline, 6 months
  Investigator administered questionnaire
Fatigue Scale for Motor and Cognitive functions (FSMC) | baseline, 3 months
  Investigator administered questionnaire
Fatigue Scale for Motor and Cognitive functions (FSMC) | baseline, 6 months
  Investigator administered questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Gobbi, MD, Principal Investigator — Neurocenter of Southern Switzerland; Claudio Gobbi, MD, Study Director — Neurocenter of Southern Switzerland
Locations (1):
- Osepdale Civico, Lugano, Canton Ticino, Switzerland

REFERENCES:
- [Background] Sellebjerg F, Barnes D, Filippini G, Midgard R, Montalban X, Rieckmann P, Selmaj K, Visser LH, Sorensen PS; EFNS Task Force on Treatment of Multiple Sclerosis Relapses. EFNS guideline on treatment of multiple sclerosis relapses: report of an EFNS task force on treatment of multiple sclerosis relapses. Eur J Neurol. 2005 Dec;12(12):939-46. doi: 10.1111/j.1468-1331.2005.01352.x. PMID 16324087
- [Background] Burton JM, O'Connor PW, Hohol M, Beyene J. Oral versus intravenous steroids for treatment of relapses in multiple sclerosis. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD006921. doi: 10.1002/14651858.CD006921.pub2. PMID 19588409
- [Background] Martinelli V, Rocca MA, Annovazzi P, Pulizzi A, Rodegher M, Martinelli Boneschi F, Scotti R, Falini A, Sormani MP, Comi G, Filippi M. A short-term randomized MRI study of high-dose oral vs intravenous methylprednisolone in MS. Neurology. 2009 Dec 1;73(22):1842-8. doi: 10.1212/WNL.0b013e3181c3fd5b. PMID 19949030
- [Background] Perumal JS, Caon C, Hreha S, Zabad R, Tselis A, Lisak R, Khan O. Oral prednisone taper following intravenous steroids fails to improve disability or recovery from relapses in multiple sclerosis. Eur J Neurol. 2008 Jul;15(7):677-80. doi: 10.1111/j.1468-1331.2008.02146.x. Epub 2008 May 6. PMID 18459972
- See also: Related information to the institution — http://www.eoc.ch/
- See also: Non profit organisazion that supports multiple sclerosis patients — http://www.multiplesklerose.ch/